CLINICAL TRIAL: NCT03412942
Title: ELITE Registry: EndovascuLar RegIstry Evaluating SafeTy, Efficacy and Patient Comfort Using the FISH ExtraCellular Matrix (SIS) Closure Device
Brief Title: EndovascuLar RegIstry Evaluating SafeTy, Efficacy and Patient Comfort (ELITE)
Acronym: ELITE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Morris Innovative Incorporated (Industry)
Collaborators: Deborah Heart and Lung Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2K17-10
Record Dates: First submitted 2017-10-11; First posted 2018-01-29 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Vascular Diseases
Keywords: Comfort; Confidence; Usage outcomes
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment with FISH device (Other): Vascular closure to be performed with FISH device.
  Interventions: Device: FISH SP

INTERVENTIONS:
Device: FISH SP — The device will be used to close the femoral artery after angiogram and/or endovascular procedure.

SUMMARY:
A single-center, prospective, cohort analysis of the Femoral Introducer Sheath and Hemostasis (FISH) vascular closure device will study 100 consecutive patients on which the device will be used to close the femoral artery after angiogram and/or endovascular procedure. Study will be conducted in order to establish the level of comfort and confidence that this device provides for both patients and physician in terms of hemodynamic and usage outcomes.

DETAILED DESCRIPTION:
The learning experience of new medical device technologies is a well-defined event but varies widely by device and user. Several factors influence rate of learning, including the device, the patient population the training technique, clear communication, and the rate of usage. Previous publication have reported on the learning curve of vascular closure technologies including; AngioSeal, Perclose & StarClose. These reports established the curve to be close to 50 experiences in order to provide predictable results.

Many prior studies have studied the safety and efficacy of vascular closure devices. However, it is substantial to also study device success when in the hands of one specific operator. This study will examine 100 consecutive subjects which the FISH vascular closure device will be used on, and examine outcomes in the following way:

Primary Endpoint:

o Safety: Severe adverse events rate (SAE) (Device related only) (transfusion/vessel occlusion)

Secondary Endpoints:

* Safety: minor adverse event rate (MAE) (Hematoma)
* Success rate (Time to Hemostasis (TTH) < 10min)
* Time to Hemostasis (TTH) mm:ss - measured from sheath pull to absence of arterial bleeding.
* Time to Ambulation (TTA) hh:mm - measured form sheath pull to walking 20 feet.
* Patient comfort - subjective measure (see scale below) measured baseline (pre-procedure/ post procedure/ 15 days and 30 days)
* Physician Confidence and Comfort (C&C)(measured every 10 patients)

ELIGIBILITY:
Inclusion Criteria:

* All patients on which a FISH device will be used for vascular closure, deemed appropriate by the Principal Investigator.

Exclusion Criteria:

* Patients on which a FISH device will not be used for vascular closure and another method will be used - deemed appropriate by the Principal Investigator (i.e. manual compressions, PerClose, AngioSeal, etc.).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Safety Questionnaire for Major Adverse Events | 30 day follow-up after device used.
  Documentation of severe adverse event related to device use (transfusion/vessel occlusion)

SECONDARY OUTCOMES:
Safety Questionnaire for Minor Adverse Events | 30 day follow-up after device used.
  Documentation of minor adverse event rate related to device use (hematoma)
Questionnaire Recording Success Rate | Within 24 hours
  Recording of time to hemostasis. TTH < 10 min will signify success
Questionnaire Measuring Time to Hemostasis (TTH) | Within 24 hours
  Documentation of time measured from sheath pull to absence of arterial bleeding in minutes:seconds
Questionnaire Measuring Time to Ambulation (TTA) | Within 24 hours
  Documentation of time measured form sheath pull to walking 20 feet in minutes:seconds
Questionnaire for Patient Comfort | Within 30 days of device
  Subjective measure, measured baseline (pre-procedure/ post procedure/ 15 days and 30 days)
Questionnaire for Physician Confidence | Within 30 days of device use
  Measured every 10 patients

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kovach, MD, Principal Investigator — Physician
Locations (3):
- United States (3):
  - Florida Research Network, LLC, Gainesville, Florida
  - Healient Physician Group, Leawood, Kansas
  - North Memorial, Robbinsdale, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided